CLINICAL TRIAL: NCT00768469
Title: A Phase 1 Study Of Neratinib (HKI-272) In Combination With Paclitaxel In Subjects With Solid Tumors
Brief Title: Study Evaluating Safety And Tolerability, Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A2-1115 / B1891001
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: HKI-272; Paclitaxel; Combination; Solid Tumor
MeSH Terms: interventions — neratinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nera 160 + Pac (Experimental): Neratinib 160 mg + Paclitaxel 80 mg/m^2
  Interventions: Drug: Neratinib; Drug: Paclitaxel
- Nera 240 + Pac (Experimental): Neratinib 240 mg + Paclitaxel 80 mg/m^2
  Interventions: Drug: Neratinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Neratinib — Administered orally, continuous, once daily.
  Other Names: HKI-272
Drug: Paclitaxel — Administered IV, on days 1, 8, 15 of 28 day cycle.

SUMMARY:
This is an open-label, phase 1 study of ascending multiple oral doses of HKI-272 in combination with paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have confirmed pathologic diagnosis of a solid tumor that is not curable with available therapy for which HKI-272 plus paclitaxel is a reasonable treatment option.
* At least 1 measurable lesion as defined by RECIST criteria.
* Eastern Cooperative Oncology Group (ECOG) 0 to 1
* LVEF within institutional limits of normal (by MUGA or ECHO).
* Screening laboratory values within the following parameters:

  * ANC: greater than or equal to 1.5 x 10E9 /L (1,500 /mm3)
  * Platelet count: 10 x 10E10 /L (100,000 /mm3)
  * Hemoglobin: greater than or equal to 9.0 g/dL
  * Serum creatinine: less than or equal to 1.5 x upper limit of normal (ULN)
  * Total bilirubin: less than or equal to 1.5 xULN · AST and ALT: less than or equal to 2.5 xULN (less than or equal to 5 x ULN if liver metastases are present)
* For women of child bearing potential, a negative urine or serum pregnancy test result before study entry. A woman of childbearing potential is one who is biologically capable of becoming pregnant. This includes women who are using contraceptives or other means of birth control or whose sexual partners are either sterile or using contraceptives.
* All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 28 days after the last dose of test article.

Exclusion Criteria:

* Prior treatment with anthracyclines with a cumulative dose of doxorubicin of greater than 400 mg/m^2, epirubicin dose of greater than 800 mg/m^2, or the equivalent dose for other anthracyclines or derivatives.
* Major surgery, chemotherapy, radical (curative intent) radiotherapy, investigational agents, or other cancer therapy within 2 weeks of treatment day 1 or non-recovery from all clinically significant acute adverse effects of prior therapies (excluding alopecia).
* Subjects with bone or skin as the only site of disease.
* Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (subjects with a history of CNS metastases or cord compression are allowable if they have been definitively treated and have been clinically stable for at least three months, and off steroids or anticonvulsants, before first dose of test article).
* QTc interval greater than 0.47 second or known history of QTc prolongation or Torsade de Pointes (TdP).
* Known hypersensitivity to paclitaxel or Cremophor EL (polyoxyethylated castor oil).
* Pregnant or breast feeding women.
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade greater than or equal to 2 diarrhea of any etiology at baseline).
* Inability or unwillingness to swallow the HKI-272.
* Treatment with a taxane within 3 months of treatment day 1.
* Pre-existing grade 2 or greater motor or sensory neuropathy.
* Any other cancer within 5 years prior to screening with the exception of contralateral breast carcinoma, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.
* Presence of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association [NYHA] functional classification of greater than or equal to 2), angina requiring treatment, myocardial infarction within the past 12 months, or any clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
* Evidence of significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, make the subject inappropriate for this study. Examples include, but are not limited to, serious active infection (ie, requiring intravenous antibiotic or antiviral agent), uncontrolled major seizure disorder, or significant pulmonary disorder (e.g. interstitial pneumonitis, pulmonary hypertension).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (2):
- Japan (2):
  - Investigational Site, Shizuoka
  - Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Started | 3 | 7
Completed | 0 | 0
Not Completed | 3 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Disease Progression | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Nera 160 + Pac | Nera 240 + Pac | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.67 (10.12) | 53.14 (8.07) | 52.10 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) - Percentage of Participants With DLT Events
Description: The incidence of DLTs in subjects with advanced solid tumors, treated with neratinib in combination with paclitaxel 80 mg/m^2. DLT was defined as any neratinib plus paclitaxel related Grade 3 or 4 nonhematologic toxicity or Grade 4 hematologic toxicity with few exceptions.
Time Frame: From first dose day through day 28.
Population: Patients with at least one dose of neratinib.
Measure: Number; unit: percentage of participants.
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Number analyzed (Participants) | 3 | 7
percentage of participants. | 0 | 0

2. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with partial response (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression/death or last tumor assessment, up to 78 weeks.
Population: Subjects who met the eligibility criteria, received at least 2 weeks of neratinib and at least 2 doses of paclitaxel, and underwent at least 1 follow-up tumor assessment at approximately cycle 2 (week 8). In the case of disease progression prior to week 8, a clinical assessment of progressive disease (PD) was adequate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Number analyzed (Participants) | 3 | 6
percentage of participants | 33.3 [0.80 to 90.6] | 50.0 [11.8 to 88.2]

3. Secondary Outcome: Progression Free Survival
Description: Number of weeks between the date of the first dose of test article and the first date of disease recurrence or progression, or death due to any cause, was documented, censored at the last evaluation, investigator assessment. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (v1.0), as at least a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as reference the nadir LD, meaning the smallest sum of the LDs recorded since the treatment started; or unequivocal progression of existing nontarget lesions; or the appearance of any new lesions.
Time Frame: From first dose date to progression/death, up to 78 weeks.
Population: Subjects who met the eligibility criteria, received at least 2 weeks of neratinib and at least 2 doses of paclitaxel, and underwent at least 1 follow-up tumor assessment at approximately cycle 2 (week 8). In the case of disease progression prior to week 8, a clinical assessment of progressive disease was adequate.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Number analyzed (Participants) | 3 | 6
weeks | 15.9 [8.4 to 78.1] | 37.1 [24.4 to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Duration of Response
Description: Number of weeks from the time at which measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever status is recorded first) until the first date on which recurrence or progressive disease (PD) is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started, for responders only, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: CR, disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From start date of response to first disease progression, up to 71 weeks.
Population: Patients with Partial Response (PR) or Complete Response (CR) in the evaluable population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Number analyzed (Participants) | 1 | 3
weeks | 70.1 [NA to NA] — Insufficient number of participants with events. | 33.1 [25.1 to NA] — Insufficient number of participants with events.

5. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose of neratinib, as determined by the incidence of DLTs, in combination with paclitaxel 80 mg/m^2, in subjects with advanced solid tumors.
Time Frame: From first dose day through day 28.
Population: Patients with at least one dose of neratinib.
Measure: Number; unit: mg
Groups:
- Nera + Pac: Neratinib + Paclitaxel 80 mg/m^2
Arm/Group | Nera + Pac
Number analyzed (Participants) | 10
mg | 240

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 28 days, up to 78 weeks.
Description: Safety Population
Arm/Group | Nera 160 + Pac | Nera 240 + Pac
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nera 160 + Pac (N=3) | Nera 240 + Pac (N=7)
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nera 160 + Pac (N=3) | Nera 240 + Pac (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 1 | 3
Catheter site pain (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 7
Influenza like illness (General disorders) | 2 | 2
Injection site reaction (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Adenoiditis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 2
Fungal skin infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2
Electrocardiogram abnormal (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 6
Somnolence (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 3
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less